CLINICAL TRIAL: NCT00268710
Title: Multicenter Phase II Study of Taxotere (Docetaxel) Administered Weekly or Every Three Weeks in Combination With Prednisone as Second Line Chemotherapy in Patients With Hormone Refractory Prostate Cancer (HRPC)
Brief Title: Docetaxel in Hormone Refractory Prostate Cancer (HRPC)[Weekly or 3weekly TAX + Prednisone in HRPC]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Canadian Urologic Oncology Group (Other)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976J_2503
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
Primary objectives:

* To determine the response rate, measurable and non measurable, to Taxotere® in the second line setting.

Secondary objectives:

* To evaluate the overall safety and toxicity of Taxotere®/prednisone combination as second line therapy in HRPC
* To evaluate PSA response (PSA: Prostate Specific Antigen)
* To evaluate symptomatic response
* To evaluate Quality of life
* To evaluate patient safety of weekly versus q3 weekly regimens of Taxotere®.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically proven prostate adenocarcinoma
* Progression or non response with previous chemotherapy regimen (excluding Taxotere®)
* Received previous mitoxantrone/prednisone or one other chemotherapy regimen including emcyt +/- vinblastine
* Castration levels of testosterone (<50 ng/dL )
* ECOG performance status 0-2
* Laboratory requirements :

  1. Hematology:

     * Neutrophils ≥ 1.5 x 10^9/L
     * Hemoglobin > 10 g/dL (prior transfusion permitted).
     * Platelets ≥ 100 x 10^9/L
  2. Hepatic function:

     * Total bilirubin < the upper-normal limit of the institution.
     * ALAT (SGPT) and ASAT (SGOT) ≤ 1.5 times the upper-normal limit of the institution.
  3. Renal function:

     * Creatinine ≤1.5 times the upper normal limit (i.e., NCI grade ≤1)
* No severe or uncontrolled disease

Exclusion Criteria

* Chemotherapy within the last 4 weeks
* Anti-androgen therapy within the last 4 weeks.
* Prior malignancy except the following: adequately treated non-melanomatous skin cancer and superficial bladder cancer from which the patient has been disease-free for >2 years.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study screening.
* Treatment with any other anti-cancer therapy (except LHRH agonists) including any prescribed compounds and/or OTC products for the treatment of prostate cancer must be stopped prior to study entry.
* Other serious illness, psychiatric or medical condition that would not permit the patient to be managed according to the protocol including active uncontrolled infection and significant cardiac dysfunction.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Pain (pain progression evaluated with the Present Pain Intensity scale form McGill-Melzack questionnaire) | During the Study Conduct

SECONDARY OUTCOMES:
Analgesics (assessed by Pain Medication Log) | During the study conduct
PSA (PSA response and PSA progression | During the study conduct
Tumor lesion assessment, | During the study conduct
Overall survival | During the study conduct
Progression-free survival | During the study conduct
Treatment emergent adverse events recorded by the investigator where intensity was according to NCI-CTC criteria: Standard hematology, blood chemistry and clinical exams. | from the inform consent signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Monique Furlan, Study Director — Sanofi